CLINICAL TRIAL: NCT03962270
Title: Effect of Extracorporeal Shock Wave in the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Mouwang Zhou, senior professional post, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2018089
Record Dates: First submitted 2018-10-30; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Knee Osteoarthritis; Cartilage Injury
Keywords: Extracorporeal Shock Wave Therapy; Knee Osteoarthritis; Cartilage Injury
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Device: shock wave device
- Control group (Sham Comparator)
  Interventions: Device: shock wave device

INTERVENTIONS:
Device: shock wave device — The experimental group (group ESWT) guided by ultrasound: conventional rehabilitation training is given priority to with strength training, application of pain when necessary, under the guidance of ultrasound ESWT treatment control group (routine rehabilitation group) : conventional rehabilitation training is given priority to with strength training, oral pain when necessary, under the guidance of ultrasound ESWT treatment (shock energy flow density of 0)

SUMMARY:
In this study, the effectiveness of ESWT in the treatment of knee OA was investigated from the perspective of cartilage injury，and to prove that shockwave could delay the early and middle stage OA progression by improving cartilage condition

ELIGIBILITY:
Inclusion Criteria:

* Knee joint ROM normal or near normal: flexion 110 ° or reach 0 ° or less
* MR prompt exist cartilage damage, there is no lack of full-thickness cartilage
* Kellgren - Lawrence (K - L) grade II - III grade
* The international association of cartilage repair cartilage damage grading system (ICRS) class I - III
* Informed consent and sign relevant documents
* Follow doctor's instructions and follow up on time

Exclusion Criteria:

* Metabolic arthritis
* Trauma of bone joint
* Inflammatory diseases
* Previous knee surgery history
* History of knee cavity injection in the past 6 months
* Serious cardiovascular diseases, pulmonary diseases or other serious diseases affecting survival, etc

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
magnetic resonance imaging of knee | Baseline (before treatment)
  t2 mapping
magnetic resonance imaging of knee | Three months after treatment
  t2 mapping

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univercity Third Hospital, Beijing, No State Or Province, China

IPD SHARING:
Plan to Share IPD: Undecided